CLINICAL TRIAL: NCT01396629
Title: Clinical Evaluation of a New Cartridge for the Implantation of Foldable Intraocular Lenses
Status: Completed | Type: Observational
Sponsor: Aurolab (Other)
Responsible Party: Sponsor
Other Study IDs: 8PN1011155
Record Dates: First submitted 2011-07-14; First posted 2011-07-19 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Cataract
Keywords: cartridge IOL
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- single group: the intra ocular lenses will be loaded in the cartridge.
  Interventions: Procedure: cartridge

INTERVENTIONS:
Procedure: cartridge — IOL cartridge coated with polymer material may ensure smooth delivery of IOL during cataract surgery

SUMMARY:
The aim of the study is to evaluate the safety and effectiveness of a new cartridge for the implantation of foldable intraocular lenses.

DETAILED DESCRIPTION:
Intraocular Lenses (IOL) Cartridge is made up of polypropylene material with coating. This cartridge is used as lens delivery system for foldable lens implantation while doing cataract surgery. The coating is made up of medical grade polyurethane and biocompatible. This coating would be useful for smooth delivery of intraocular lens.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 60
* Senile cataract
* Nuclear Sclerosis grade I and grade II

Exclusion Criteria:

* Inherent zonular weakness
* Shallow anterior chamber
* PXF
* Traumatic cataract
* Uveitis and Complicated cataract
* Dense PSCC and PPC

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patient with senile cataract or Nuclear Sclerosis grade I and grade II and age between 40-60
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2011-07; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
intra operative complication | post operative day 1
  to asssess the incidence of cartridge related post operative complications occurring in the anterior chamber on day 1

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Haripriya Aravind, MBBS., MS.,, Principal Investigator — HOD of IOL & Cataract clinic, Aravind Eye Hospital, Madurai
Locations (1):
- Aravind Eye Hospital, Madurai, Tamil Nadu, India